CLINICAL TRIAL: NCT04032600
Title: Malignant Ascites in Ovarian Cancer: Impact of Total Paracentesis on Hemodynamics
Acronym: ATLANTIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Dr. Klaus Pietzner, Principal Investigator, Consultant of Gynaecological Oncology, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EA 1/224/16
Record Dates: First submitted 2018-02-11; First posted 2019-07-25 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2019-07

CONDITIONS: Malignant Ascites; Ovarian Cancer; Hemodynamic Instability
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Paracentesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full paracentesis (Other): All ascites is drained
  Interventions: Procedure: Paracentesis
- Fractioned paracentesis (Other): 3 Liters are drained, then the drain is clamped and the rest of the ascites is drained on the next day
  Interventions: Procedure: Paracentesis

INTERVENTIONS:
Procedure: Paracentesis — Full versus partial paracentesis (3 liters)

SUMMARY:
The ATLANTIS-study was designed to determine the safety of a full paracentesis in patients with malignant ascites due to ovarian cancer. The underlying hypothesis states, that full paracentesis does not impair safety, compared to fractioned paracentesis with clamping of the drain. Half of the patients will receive a full paracentesis, while the other half will receive fractioned paracentesis with clamping of the drain after 3 liters of ascites was evacuated. All patients receive extensive monitoring of hemodynamics and kidney function.

DETAILED DESCRIPTION:
Background: Malignant ascites is common in ovarian cancer and often causes symptoms such as abdominal pressure and shortness of breath, resulting in an decreased quality of life for the patient. Paracentesis is a safe and easy method for symptom relief. But no guidelines exist on the management of ascites drainage in ovarian cancer. In many cases a partial paracentesis is performed, due to fear of hemodynamic instability or kidney failure, with partial drainage of the intraperitoneal fluid on the first day and subsequent drainage on the next day. As there is no study that reported a deteriorated health due to full paracentesis in ovarian cancer, the decision whether a partial or total paracentesis is performed depends entirely on the department or the physician.

Since a total paracentesis can be performed as an out-patient treatment, this approach is often preferred by the patient. Full paracentesis is also more efficient and cost-effective.

The objective of the ATLANTIS-study is to prove the safety of total paracentesis regarding hemodynamic changes and kidney failure.

Methods: ATLANTIS is a randomized, prospective, clinical study that aims to include 60 patients. Patients with histologically confirmed epithelial ovarian, fallopian tube and peritoneal cancer are randomized into two arms: Partial (3 Liter) and total paracentesis. Before, during and for two hours after the paracentesis, an advanced hemodynamic monitoring is performed to ensure the patients' safety. The monitoring includes mean arterial pressure and stroke volume. After the initial phase of extensive monitoring (2 hours), the blood pressure is measured for a period of 24 hours to evaluate not only short term, but also long-term hemodynamic changes. Before and 24 hours after the paracentesis, blood samples are analyzed to detect a potential acute kidney failure.

ELIGIBILITY:
Inclusion criteria:

* Histologically confirmed ovarian cancer, peritoneal cancer or fallopian tube cancer
* Symptomatic (e.g. abdominal pressure, pain, shortness of breath) malignant ascites with clinical indication for paracentesis and sonographic estimate of >3 liters
* Patient information and written informed consent

Exclusion criteria:

* Age <18 years
* Missing written informed consent
* Lack of sufficient knowledge of german or english language
* No willingness to consent to the storage or distribution of anonymised disease-specific data inside the clinical trial
* Placement inside a state facility due to judicial order
* Employee status at Charite-University Medicine of Berlin
* Chronic kidney insufficiency defined as serum creatinin levels >1,2 g/dl at time point of admission
* Active neurologic/psychiatric disorder at time point of admission
* Cardiac insufficiency defined as >NYHA I at time point of admission
* Manifest ileus at time point of admission
* Manifest chronic arterial hypo- or hypertension, defined as chronic baseline systolic pressure of <90 or >140 mmHg and diastolic pressure of <70 and >90 mmHg
* Active infection
* Blood clotting disorder (congenital or acquired)
* Thrombocytopenia (platelets <80 000/nl)
* Active participation in another clinical intervention trial at time point of admission
* Chronic atrial fibrillation on time point of admission
* Status post cardiac pacer implantation
* Liver cirrhosis
* Liver metastases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2019-09-09 (Actual)

PRIMARY OUTCOMES:
Change of stroke volume | 20 minutes prior to paracentesis, during paracentesis up to the end of paracentesis, an average of 50 minutes
  Stroke volume is measured by advanced hemodynamic monitoring
Change of mean arterial pressure | 20 minutes prior to paracentesis, during paracentesis up to the end of paracentesis, an average of 50 minutes
  Mean arterial pressure is measured by advanced hemodynamic monitoring

SECONDARY OUTCOMES:
Incidence of side effects in the post-paracentesis interval | 24 hours after the finish of the paracentesis
  Incidence of hypotension (medical intervention indicated) and impairment of kidney function (KIDIGO criteria)
Incidence of symptoms in the post-paracentesis interval | 24 hours after the finish of the paracentesis
  Incidence of hypotension (medical intervention indicated) and impairment of kidney function (KIDIGO criteria)
Change of stroke volume in the post-paracentesis interval | 2 hours after the finish of the paracentesis
  Stroke volume is measured by advanced hemodynamic monitoring
Change of mean arterial pressure in the post-paracentesis interval | 2 hours after the finish of the paracentesis
  Mean arterial pressure is measured by advanced hemodynamic monitoring
Change of laboratory values | Serial measurements: 2 hours prior to paracentesis, 24 hours after paracentesis
  Measurement in plasma (Blood count, creatinin, AST, ALT, urea, aldosterone, renin, sodium, potassium, albumin, C-reactive protein, leukocytes)
Urine excretion | 24 hours after the finish of paracentesis
  Urin volume
Quality of life- pre and post paracentesis: EQ-5D questionnaire | 2 hours before paracentesis, 24 hours after paracentesis and 1 week after paracentesis
  Measured with the EuroQuol-Group 5 Dimensions - Visual analog scale (EQ-5D VAS) questionnaire, the questionnaire directs to characterize the quality of life by mobility, activities, pain and fear and subjective scale between 1 (worst) and 100 (best)
Ascites related symptoms- pre and post paracentesis | 2 hs before paracentesis, 24-hours after paracentesis and 1 week after paracentesis
  Measured with the and Functional Assessment of Chronic Illness Therapy-Ascites Index (FACIT-AI) questionnaire, the questionnaire directs to characterise the symptoms associated to ascites regarding 13 factors e.g. appetite, sleep, activities, symptoms, emotional distress by 0 to 4 points. The maximum score is 52 (best result: 13x4), 0 is the minimum score (worst result 13x0)
Measurement of exact drainage volume | Within 1 hour after the finish of paracentesis
  Measurement of exact drainage volume in millilitre
VEGF (vascular endothelial growth factor) level | Within 1 hour after the finish of paracentesis
  Measurement of the concentration of hormone vascular endothelial growth factor in ascites
Change of venous return and mean systemic filling pressure | 20 minutes prior to paracentesis, during paracentesis up to the end of paracentesis, an average of 50 minutes
  Venous return and mean systemic filling pressure is measured by advanced hemodynamic monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Pietzner, MD, Principal Investigator — Charite-University Medicine of Berlin, Department of Gynecology
Locations (1):
- Charite-University Medicine of Berlin, Department of Gynecology-Campus Virchow Klinikum, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided